CLINICAL TRIAL: NCT00653731
Title: Testing Three Interventions for Clinical Effectiveness in Long Term Care Residents With Dementia: Snoezelen, Structured Reminiscence Therapy, 10-minutes Activation. A Cluster-randomized Controlled Trial.
Brief Title: Effective Strategies for Dementia Care
Acronym: WISDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Johann Behrens, Professor, Martin-Luther-Universität Halle-Wittenberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PfVMS-T6
Record Dates: First submitted 2008-04-02; First posted 2008-04-07 (Estimated); Last update posted 2011-08-31 (Estimated); Status verified 2011-08

CONDITIONS: Dementia; Cognitive Impairment
Keywords: dementia; snoezelen; structured reminiscence therapy; 10-minutes activation; apathy
MeSH Terms: conditions — Dementia; Cognitive Dysfunction; Lethargy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Snoezelen © (Experimental)
  Interventions: Behavioral: Snoezelen ©
- Reminiscence (Experimental)
  Interventions: Behavioral: structured reminiscence therapy
- 10 min activation (Experimental)
  Interventions: Behavioral: 10-minutes activation
- Talk (Active Comparator)
  Interventions: Behavioral: Unstructured verbal communication

INTERVENTIONS:
Behavioral: Snoezelen © — Nursing individual intervention one time a week for 20 minutes
  Arms: Snoezelen ©
Behavioral: structured reminiscence therapy — Individual nursing intervention: one time a week 20 minutes
  Arms: Reminiscence
Behavioral: 10-minutes activation — Individual nursing intervention: two times a week for 10 minutes
  Arms: 10 min activation
Behavioral: Unstructured verbal communication — Individual nursing intervention: one time a week for 20 minutes
  Arms: Talk

SUMMARY:
The purpose of this study is to determine whether the interventions of Snoezelen, structured reminiscence therapy and 10-minutes activation are effective to reduce apathy in long term care residents with dementia.

DETAILED DESCRIPTION:
Design:

Cluster-randomized controlled trial with 20 nursing homes in Saxony and Saxony-Anhalt (Germany).

ELIGIBILITY:
Inclusion Criteria:

* Dementia
* Informed consent by legal guardian
* MMSE ≤ 24

Exclusion Criteria:

* Korsakoff's syndrome
* Age ≤ 55 years
* Cognitive impairment other cause than dementia

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 327 (Actual)
Dates: Start 2008-02; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Apathy Evaluation Scale (Marin et al. 1991) | 12 months

SECONDARY OUTCOMES:
Neuropsychiatric Inventory (Cummings 1997) | 3, 6 and 12 months
Apathy Evaluation Scale (Marin et al. 1991) | 3 and 6 months
Staff Observation Aggression Scale (Nijman et al. 1997) | 3,6 and 12 months
Nottingham Health Profile (Bureau-Chalot et al. 2002) staff-related measurement | 6 and 12 months
Smiley Analogue Scale for Well-Being | 3, 6 and 12 months
PASTA (Zimber 2001) staff-related measurement | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Johann Behrens, PhD, Principal Investigator — Martin-Luther-University Halle-Wittenberg
Locations (1):
- Institut für Gesundheits- und Pflegewissenschaft, Medizinische Fakultät, Martin-Luther-Universität Halle-Wittenberg, Halle, SAN, Germany

REFERENCES:
- [Derived] Berg A, Sadowski K, Beyrodt M, Hanns S, Zimmermann M, Langer G, Becker C, Lautenschlager C, Behrens J. Snoezelen, structured reminiscence therapy and 10-minutes activation in long term care residents with dementia (WISDE): study protocol of a cluster randomized controlled trial. BMC Geriatr. 2010 Jan 31;10:5. doi: 10.1186/1471-2318-10-5. PMID 20113526